CLINICAL TRIAL: NCT04814082
Title: Prospective Functional, Gait, and Outcome Comparison Study of Medial Pivot
Brief Title: Prospective Functional, Gait, and Outcome Comparison Study of Medial Pivot Versus Single Radius Design for Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LifeBridge Health (Other)
Collaborators: Rubin Institute for Advanced Orthopedics (Unknown); MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1679091
Record Dates: First submitted 2021-02-03; First posted 2021-03-24 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Knee; Knee Osteoarthritis; Osteoarthritis Knees Both; Osteoarthritis Knee Left; Osteoarthritis Knee Right; Knee Pain Chronic; Knee Disease; Arthropathy of Knee Joint
Keywords: Total Knee Arthroplasty; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Medial-Pivot Knee System (Active Comparator): Total Knee Arthroplasty will be done by implanting the MicroPort Medial Pivot Knee System into subjects.
  Interventions: Device: MicroPort Evolution Medial-Pivot Knee System (Cruciate-substituting)
- Single Radius Design Total Knee System (Active Comparator): Total Knee Arthroplasty will be done by implanting the Stryker Triathlon Tritanium Knee System into subjects.
  Interventions: Device: Stryker Triathlon Tritanium Knee System (Condylar Stabilizing)

INTERVENTIONS:
Device: MicroPort Evolution Medial-Pivot Knee System (Cruciate-substituting) — Medial Pivot Knee System
  Arms: Medial-Pivot Knee System
Device: Stryker Triathlon Tritanium Knee System (Condylar Stabilizing) — Single Radius Design Total Knee System
  Arms: Single Radius Design Total Knee System

SUMMARY:
Patients with degenerative joint disease can effectively be treated with a primary total knee replacement to reduce pain and improve function in their daily lives. Theoretically, achievement of normal knee motion using a medial pivot design in total knee replacements can be recreated in comparison to single radius designs, which could lead to an improvement in post-surgical outcomes and satisfaction with the procedure. The aim of this study is to compare two types of implant designs (medial pivot and single radius) in a total knee replacement using clinical outcomes, patient reported outcomes, and overall function assessed by a specialized gait laboratory.

DETAILED DESCRIPTION:
This is a single center, cohort study in 100 adult subjects undergoing primary total knee arthroplasty that will receive one of the two total knee device systems.

Primary total knee replacement is an effective treatment for relieving pain and improving function for patients with degenerative joint disease. Recently, design of knee implants in a total knee replacement have received increased interest, particularly the medial pivot designs. Single-radius implants are designed to minimize instability throughout the functional range of movement. Medial pivot total knee designs theoretically recreate more normal knee motion when compared to single radius designs. Both implant designs are commonly used for total knee replacements. Outcomes of TKA are evaluated by multiple methods including implant/device survivorship, radiographic assessments, clinical examinations, and patient reported outcome measures (PROMS). Laboratory based gait analysis performed at a specialized research facility is not commonly conducted in patients with positive outcomes post-surgery as this is associated with high cost. There is currently not enough research comparing these two designs directly. Research is required to determine which design may provide better clinical outcomes and satisfaction with the procedure.

In addition to your normal standard clinical care, there will be scheduled pre-operative, operative, 6-week, 6 month, 12 month, 24 month, 36 month, and 60 month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or non-pregnant female aged between 18 and 75 years of age.
* Subject is willing to provide informed consent to participate in the research study.
* Subject is indicated for a primary total knee arthroplasty (TKA) based on the approved labeling of knee implant, either a medial pivot or single radius design, specifically: MicroPort Evolution Medial-Pivot Knee System, Cruciate Retaining (CS) or Stryker Triathlon Tritanium (CS)
* Subject does not have a history of previous prosthetic replacement device on the operative knee.
* Subject is currently ambulating and does not have a condition on the contralateral limb in the opinion of the investigator that would interfere with the gait laboratory evaluations.
* Subject is willing and able to comply with the schedule of events for the study and is available to return to the clinic for all required follow-up visits.

Exclusion Criteria:

* Subject has a Body Mass Index (BMI) >40
* Subject has a diagnosis of avascular necrosis or inflammatory arthritis.
* Subject has any mental or neuromuscular disorder that would create an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* Subject is a prisoner
* Subject has any condition, in the opinion of the Investigator that might interfere with the evaluation of the study objectives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Mechanics | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  Knee flexion/extension, varus/valgus, and internal/external rotation will be measured (in degrees) and analyzed using the KneeKG system during incline and decline walking.
Change in Anterior/Posterior Knee Translation | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  This parameter will be measured (in mm) and analyzed using the KneeKG system during incline and decline walking.
Change in Initial Peak Loading Force | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  This parameter will be measured (in N) and analyzed using the KneeKG system during normal walking.
Change in Active and Passive Range of Motion | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  Active and passive range of motion will be measured (in degrees) using a goniometer.
Change in Quadriceps Lag | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  Quadriceps lag will be measured (in degrees) in both the sitting and supine positions.
Change in Timed up and Go Test (TUG) | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  This parameter will be measured in seconds and requires a patient to rise from a chair walk three meters and return to the chair again as quickly as possible.
Change in Five Times Sit to Stand Test | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  This parameter will be measured in seconds and will collect the amount of time it takes a patient to transfer from a seated to a standing position and back to sitting five times.
Change in Single Limb Stance Test for Both Knees | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  This parameter will be measured in seconds and will collect the amount of time a patient is able to stand unassisted on one leg.
Change in Timed Ascent and Descent of One Flight of Stairs Test | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  This parameter will be measured in seconds and will collect the amount of time it takes a patient to ascend and descend one flight of stairs (8-14 steps).
Change in Quadriceps Muscle Strength | Pre-operative; Post-operative - 3 month and 12 month follow-up visit
  This parameter will be measured (in lbs/in) using a dynamometer for quadricep muscle strength assessment.

SECONDARY OUTCOMES:
Implant Survivorship | Post-operative - 6 week, 6 month, 12 month, 24 month, 36 month, and 60 month follow-up visit
  Radiographic assessment using AP and lateral knee X-rays to analyze implant position, radiolucencies, fracture, and osteolysis.
Post-surgical Complications | Operative visit; Post-operative - 6 week, 6 month, 12 month, 24 month, 36 month, and 60 month follow-up visit
  All complications related to the procedure will be documented.
Evidence of Osteolysis | Pre-operative; Post-operative - 6 week, 6 month, 12 month, 24 month, 36 month, and 60 month follow-up visit
  X-rays will be evaluated to look for presence of a radiolucent area, especially > 2mm, around implant or cement with sclerotic border.
Change in Knee Society Score (KSS) Short Form | Pre-operative; Post-operative - 6 week, 6 month, 12 month, 24 month, 36 month, and 60 month follow-up visit
  25 question items assessing symptoms, patient satisfaction, patient expectation, and their level of functional activity of their knee. Scores range from 0-100 with higher scores representing better outcomes.
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre-operative; Post-operative - 6 week, 6 month, 12 month, 24 month, 36 month, and 60 month follow-up visit
  42 question items assessing a patient's opinion about their health, symptoms, and function of their knee. Scores range from 0-100 with zero representing severe knee problems and 100 indicating no knee problems.
Change in Patient Reported Outcomes Measurement Information System (PROMIS-10) | Pre-operative; Post-operative - 6 week, 6 month, 12 month, 24 month, 36 month, and 60 month follow-up visit
  10 question items assessing overall physical, mental, and social health of the patient. Each question item is scored separately on 1-5 scale and total scores are combined into 2 groups - Global Physical Health Score and Global Mental Health score. A T-score is calculated with the 2 previous scores against the general population with a higher T-score representing better outcomes.
Change in Forgotten Joint Score FJS | Pre-operative; Post-operative - 6 week, 6 month, 12 month, 24 month, 36 month, and 60 month follow-up visit
  12 question items evaluating how "aware" a patient is of their operative joint during daily activities. Scores range between 0-100 with higher scores indicating a patient is able to forget the joint on a daily basis or low joint awareness.

CONTACTS AND LOCATIONS:
Overall Officials: James Nace, MD, Principal Investigator — LifeBridge Health
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States